CLINICAL TRIAL: NCT03035149
Title: Exercise Capacity and Dyspnea in Obese Patients With Metabolic Syndrome: Effects of Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Collaborators: Ontario Lung Association (Other); The Ottawa Hospital (Other)
Responsible Party: Principal Investigator, Dr. Nha Voduc, MD, University of Ottawa
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2005213-01H
Record Dates: First submitted 2017-01-24; First posted 2017-01-27 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Obesity; Metabolic Syndrome
Keywords: Obesity; Metabolic Syndrome; Dyspnea; Pulmonary Function; Exercise Capacity
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weight Management Program (Experimental): Obese subjects participate in a year long medically supervised weight management program.
  Interventions: Other: Weight Management Program
- Normal Weight Controls (No Intervention): Normal weight age and sex-matched controls. Unlike the obese subjects, the controls did not participate in the Weight Management Program. Pulmonary function, exercise performance and dyspnea results for normal weight controls were compared against the results for obese subjects.

INTERVENTIONS:
Other: Weight Management Program — Obese subjects partake in a medically supervised weight management program. This lifestyle modification program involves weekly three hour sessions for six months and monthly sessions for six months. The first twelve weeks comprise an initial weight loss phase when patients are placed on a 900 Kcal/day meal replacement. This is followed by a four week transition to a 1200-1800 Kcal diet followed by a ten week maintenance phase of 10 weekly sessions.The majority of weight loss occurs during the first 26 weeks followed by a 26 week period of stabilization of weight loss. Hence subjects are evaluated after the first 26 weeks.
  Arms: Weight Management Program

SUMMARY:
Dyspnea is a common complaint in obese patients. The mechanisms behind this dyspnea and the effects of weight loss on dyspnea are not completely understood. The objectives of this study were to examine the relationships between exercise parameters and dyspnea in obesity and assess the effects of weight loss.

The investigators compared pulmonary function, exercise performance and dyspnea in 34 patients with abdominal obesity and metabolic syndrome (MS) against 34 age and sex-matched controls. The study also assessed within-group changes in physiology and symptoms in a subset of patients following participation in a weight management program.

Because obesity is a heterogeneous condition, with variable genetic associations, co-morbidities and distributions of adipose tissue, the study focused on patients with abdominal obesity who met diagnostic criteria for metabolic syndrome.

DETAILED DESCRIPTION:
The study has two parts: first, the investigators compared dyspnea, pulmonary function and exercise measurements between obese patients and control subjects with normal weight; then, the investigators assessed the effects of medical weight loss in the obese group on these parameters. Baseline dyspnea was assessed using the baseline dyspnea index.The effect of weight loss on dyspnea was assessed using the transitional dyspnea index. The main physiologic measurement of interest was the inspiratory capacity (L, measured at rest and during exercise).

ELIGIBILITY:
Inclusion Criteria:

* Individuals accepted into the behavioural weight management program at the Ottawa Hospital Bariatric Centre
* Age between 20 and 60 years
* BMI greater than 30
* Abdominal girth (for females) greater than 88 cm
* Abdominal girth (for males) greater than 102 cm
* Plus any two of the other criteria for Metabolic Syndrome:

  i.e. Blood Pressure greater or equal to 130/85; Fasting Glucose greater or equal to 6.1 mmol/L
* Controls-normal weight (NW) and sedentary

Exclusion Criteria:

* Smoker
* Any medical conditions which would affect exercise performance
* Use of medications that could affect exercise performance (i.e. Beta-blockers)
* Inability to pedal on a cycle ergometer and provide reproducible inspiratory capacity (IC) measurements

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2005-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Dyspnea (measured by Transitional Dyspnea Index) | Within 6 months following completion of 6 months (weight loss period) in the weight management program
  Dyspnea was assessed using a questionnaire based on the Transitional Dyspnea Index
Resting Inspiratory Capacity (L) | Within 6 months following completion of 6 months (weight loss period) in the weight management program
  Inspiratory capacity (difference between total lung capacity and functional residual capacity), measured at rest
Inspiratory Capacity during Exercise (L) | Within 6 months following completion of 6 month (weight loss period) in the weight management program
  Inspiratory capacity measured at identical time points during incremental exercise tests, performed before and after weight loss

CONTACTS AND LOCATIONS:
Overall Officials: Nha Voduc, MD, Principal Investigator — University of Ottawa
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No